CLINICAL TRIAL: NCT00817141
Title: Is Urinary Catheter Necessary After Fast-Track Colonic Surgery?
Brief Title: Urinary Catheter and Fast-track Surgery
Status: Completed | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Forget Patrice, MD PhD, Université Catholique de Louvain
Other Study IDs: 2008/12MARS/82
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Urinary Complications
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Without urinary catheter
  Interventions: Other: Observational study, no intervention

INTERVENTIONS:
Other: Observational study, no intervention — Observation of the complications seen without urinary catheter (which is the habitual protocol in our institution)

SUMMARY:
Urinary catheter was placed during several days after colonic surgery. Nevertheless, it is probably unnecessary after Fast-Track colonic surgery. No prospective data permit to confirm it.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for Fast Track colonic surgery

Exclusion Criteria:

* Urinary pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for Fast Track colonic surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Incidence of urinary retention necessitating catheterisation | 72 hours

SECONDARY OUTCOMES:
Other urinary complications and modification of the Fast Track protocol | 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- St Luc Hospital, Brussels, Belgium